CLINICAL TRIAL: NCT02076659
Title: A Dose-finding, Pharmacokinetic Phase I Study of the Human Monoclonal Antibody-cytokine Fusion Protein F8IL10 (Dekavil) in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: Combination Therapy of F8IL10 and Methotrexate in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-F8IL10-02/08; 2008-008729-31 (EudraCT Number)
Record Dates: First submitted 2014-02-24; First posted 2014-03-03 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
Keywords: F8; IL10; Interleukin; monoclonal; antibody; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F8IL10 + MTX (Experimental): Ten cohorts of 3-6 RA patients will be treated at increasing doses per cohort of F8IL10 plus fixed doses of MTX and folic acid.
  An additional 12 patients will be randomized (6+6) in a double blind, placebo controlled cohort with F8IL10 given at RD and placebo. In both arms, MTX will be administered as concomitant medication.
  In all coohorts a stable dose of folic acid (5 mg) will be administered on Day 2.
  Interventions: Drug: F8IL10; Drug: Methotrexate

INTERVENTIONS:
Drug: F8IL10 — Weekly administration of F8IL10 (from 6 to 600 μg/kg), starting from 6 μg/kg cohort 1. The cohort 10 represents the last dose-level of the study.
  F8IL10 will be administered as subcutaneous (s.c.) injections. Patients will receive 4 cycles of treatment unless there is unacceptable toxicity or withdrawal of consent.
Drug: Methotrexate — Methotrexate will be administered at a fixed dose of 10-15 mg on Day 1, orally (p.o.), subcutaneously (s.c.) or intramuscularly (i.m.).
  Patients will receive 4 cycles of treatment unless there is unacceptable toxicity or withdrawal of consent.

SUMMARY:
Phase I, multicenter, open-label, dose escalation study to test the efficacy and safety of F8IL10 and methotrexate when given as a combination in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
The study is designed to explore whether F8IL10 can be safely administered in combination with standard-dose of MTX in patients with active rheumatoid arthritis and to determine the recommended dose of F8IL10 when combined with MTX.

As soon as the MTD/RD is determined, an additional 12 patients will be randomized (6+6) between F8IL10 (RD) and placebo to further investigate the safety and pharmacacodynamics profile of the study treatment.

Methotrexate (MTX) will be administered as concomitant medication in the dose escalation as well as in the randomized part of the study.

ELIGIBILITY:
Inclusion criteria

1. Patients aged ≥ 18 and < 75 years.
2. Diagnosis of RA according to ACR criteria (1987) with a disease duration exceeding 12 months.
3. Active RA (DAS28 ≥ 3.2) for ≥ 4 months at time of signing informed consent.
4. Receiving treatment on an outpatient basis.
5. MTX at 10-15 mg/w for a period ≥ 8 weeks prior to treatment.
6. Inadequate clinical response to at least one anti-TNF therapy applied for at least 4 months.
7. If patients are receiving an oral corticosteroid, the dose must have been stable for at least 25 out of 28 days prior to study treatment and the dose must be less than 10 mg/day (prednisolone equivalent).
8. All acute toxic effects of any prior therapy must have returned to classification "mild" according to RCTC V.2.0 [1] .
9. Sufficient hematologic, liver and renal function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin (Hb) ≥ 9.5 g/dL
   * Alkaline phosphatase (AP), alanine aminotransferase (ALT) and or aspartate aminotransferase (AST) ≤ 3 x upper limit of normal range (ULN), and total bilirubin ≤ 2.0 mg/dL (34.2 µmol/L)
   * Creatinine ≤ 1.5 ULN or 24 h creatinine clearance ≥ 50 mL/min
10. Documented negative test for human immunodeficiency virus, HBV, and HCV. For patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV DNA is required.
11. Male and female patients, who are potentially fertile, must agree to use adequate contraceptive methods at the beginning of the screening visit that must be continued until 3 months following the last treatment with study drug.
12. Negative serum pregnancy test (for women of child-bearing potential only) at screening.
13. Signed and dated Ethics Committee-approved Informed Consent Form indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the study.
14. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion criteria

1. Presence of active infections (e.g. requiring antibiotic therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or would interfere with the study objectives or conduct.
2. Pregnancy, lactation or unwillingness to use adequate contraceptive methods.
3. Active or latent tuberculosis (TB).
4. Chronic active hepatitis or active autoimmune diseases other than RA.
5. History of currently active primary or secondary immounodeficiency.
6. HIV Infection.
7. Acute or chronic-active infection with HBV or HCV, as assessed by serology or HBV DNA.
8. Evidence of active malignant disease at screening or advanced malignancies diagnosed within the previous 5 years.
9. Any previous treatment with alkylating agents, such as cyclophosphamide or chlorambucil or with total lymphoid irradiation.
10. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
11. Treatment with warfarin or other coumarin derivatives.
12. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
13. Irreversible cardiac arrhythmias requiring permanent medication.
14. Clinically significant (to clinical investigator's discretion) abnormalities in baseline MUGA, ECHO or ECG analyses.
15. Uncontrolled hypertension.
16. Ischemic peripheral vascular disease (Grade IIb-IV).
17. Severe diabetic retinopathy.
18. Major trauma including surgery within 4 weeks of administration of study treatment.
19. Known history of allergy or other intolerance to IL10, MTX, folic acid or other drugs based on human proteins/peptides/antibodies.
20. In vivo exposure to monoclonal antibodies for biological therapy (e.g., adalimumab,infliximab golimumab, tocilizumab, certolizumab pegol) less than 8 weeks prior to administration of study medication.
21. Treatment with rituximab less than 4 months prior to administration of study medication.
22. Treatment with fusion proteins (e.g. abatacept, etanercept) less than 4 weeks prior to administration of study medication.
23. Treatment with any investigational agent within the 6 weeks before study treatment.
24. Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
25. Growth factors or immunomodulatory agents, including anakinra, within 7 days of the administration of study treatment.
26. Neuropathy > Grade 1 or Neuropathies or other painful conditions (not RA-related) that might interfere with pain evaluation.
27. Patients required to be treated with corticosteroids at a dose > 10 mg/day or with immunosuppressant drugs other than MTX on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
28. History of alcohol, drug or chemical substance abuse within the 6 months prior to screening.
29. Body weight of >100 kg.
30. Any condition that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events that are related to treatment and classified as DLTs for each administered dosage | Up to day 28
  To establish the MTD and the RD of F8IL10 when administered in combination with methotrexate

SECONDARY OUTCOMES:
Maximum drug concentration [Cmax] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Time to reach maximum drug concentration [Tmax] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Terminal half-life [t1/2] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Area under the drug concentration-time curve [AUC(0 - t last)] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Area under the drug concentration-time curve, extrapolated to infinity [AUC] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Accumulation ratio for AUC [R AUC] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Accumulation ratio for Cmax [Rmax] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Accumulation ratio for Cmin [R min] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Total clearance following the dose administered [CL] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Volume of distribution at steady state [Vss] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Mean residence time [MRT] | At day 1, 4, 5, 6 of week 1; at day 1, 2, 3, 4, 5, 6 of week 4
  Pharmacokinetics assessment of F8IL10 through blood sampling
Human anti-fusion protein antibodies (HAFA) levels | 1) at day 1 of week 1; 2) at day 1 of week 4; 3) from week 5 up to week 9 (EoT visit)
  Investigate the potential induction of human anti-fusion protein antibodies (HAFA) through standard laboratory analysis.
Response rate according to EULAR criteria (Good, Moderate and Non-responders) based on DAS28 score | 1) from day -14 up to day 0 (screening); 2) at day 1 of week 5; 3) at day 1 of week 9; 4) from week 9-13 up to week 57-61, every 4 weeks (safety/efficacy follow-up)
  To explore the antiarthritic activity of the study medication in patients with active rheumatoid arthritis.
ACR 20, ACR 50, ACR 70 response rate | 1) from day -14 up to day 0 (screening); 2) at day 1 of week 5; 3) at day 1 of week 9; 4) from week 9-13 up to week 57-61, every 4 weeks (safety/efficacy follow-up)
  To explore the antiarthritic activity of the study medication in patients with active rheumatoid arthritis.
Change from baseline in DAS28 | 1) from day -14 up to day 0 (screening); 2) at day 1 of week 5; 3) at day 1 of week 9; 4) from week 9-13 up to week 57-61, every 4 weeks (safety/efficacy follow-up)
  To explore the antiarthritic activity of the study medication in patients with active rheumatoid arthritis.
Relative change over time of blood biomarkers | From day -14 up to day 0 (screening); at day 1 of week 1; at day 1 of week 5 /week 9 (EoT); from week 7 up to week 11 (safety follow-up); from week 11 up to week 15 (efficacy follow-up); from week 11-15 up to week 57-61, every 4 weeks (total follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Galeazzi, Prof, Principal Investigator — Siena University Hospital
Locations (5):
- Italy (5):
  - Policlinico San Matteo, Pavia, Pavia
  - Pisa University Hospital, Pisa
  - Azienda Ospedaliera San Camillo-Forlanini Roma, Roma
  - Policlinico A. Gemelli, Università Cattolica del Sacro Cuore, Roma
  - Siena University Hospital, Siena